CLINICAL TRIAL: NCT01963195
Title: An Open, Single Center Trial to Evaluate the Efficacy and Safety of Dose Escalation of Icotinib in Advanced NSCLC Patients After TKI Therapy
Brief Title: Evaluation of the High Dose of Icotinib in Advanced Lung Cancer Patients After Failure of Target Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, Pan Yueyin, Professor, Anhui Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DEI-ADNSCLC
Record Dates: First submitted 2012-01-04; First posted 2013-10-16 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: NSCLC
Keywords: Adverse Reaction to Drug; Self Efficacy
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — icotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Icotinib (Experimental): Patients can accept the treatment with Icotinib (250/375/500mg tid) until disease progression or unacceptable toxicity occurred. The overall study period takes about 24 months
  Interventions: Drug: Icotinib

INTERVENTIONS:
Drug: Icotinib — Patients can accept the treatment with Icotinib (250/375/500mg tid) until disease progression or unacceptable toxicities occurred. The overall study period takes about 24 months
  Other Names: high dose of Icotinib

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of dose escalation of Icotinib in advanced non small cell lung cancer (NSCLC) patients after the therapy of Icotinib, Iressa and Tarceva.

DETAILED DESCRIPTION:
* 1:to evaluate the efficacy correlation between the tyrosine kinase inhibitor (TKI) drugs and high-dose Icotonib group in advanced NSCLC patients with high -dose Icotinib going on after the routine TKI therapy
* 2 to evaluate the efficacy correlation between different high-dose group in advanced NSCLC patients with high -dose Icotinib going on after the routine TKI therapy

ELIGIBILITY:
Inclusion Criteria:

1. NSCLC patients were confirmed by histology or cytology
2. The time interval must be over 4 weeks from previous chemotherapy to registration to participate in this experiment if he or she received chemotherapy,and also have any toxicity to recover.
3. at least one measureable lesion accord to RECIST 1.1 criteria and the lesion accepted no radiotherapy.

   * 1 at least one measureable lesion .if only one measureable lesion, the biological nature must be confirmed by cytology or histology.
   * 2 a single diameter of lesion could be measured by at least one of the following methods: Chest or abdominal computed tomography(CT)or magnetic resonance imaging(MRI),conventional methods of diameter at least 20mm diameter spiral CT OR at least 10mm.
4. ECOG 0-2 score
5. at least 12 weeks of expected survival time
6. Women of childbearing age must have a pregnancy test 7 days before treatment and the result were negative ,men of childbearing age: surgical sterilization or treatment during and after the end of three months to take contraceptive measures
7. understand and sign a written informed consent voluntarily.

Exclusion Criteria:

If the subject meet any of the following exclusion criteria ,he is no eligible to participate in this study,

1. Before enrollment in this trial have used Erbitux, Herceptin and carried out anti-cancer therapy.
2. use of phenytoin, carbamazepine, rifampicin, phenobarbital or St. John's Wort when take this trial
3. severe allergies to Icotinib

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-02; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
safety and efficacy | 2 years
  1. The efficacy of dose escalation of Icotinib in advanced NSCLC patients after failure of TKI (Icotinib 125mg po tid. Iressa 250mg po qd. Tarceva 150mg po qd) therapy will be evaluated according to the revised RECIST 1.1 (Response Evaluation Criteria In Solid Tumors).
  2. The safety of high dosage of Icotinib will be evaluated according to the Common Terminology Criteria for Adverse Events (CTCAE) v4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Yueyin Pan, MD, Principal Investigator — Anhui Medical University
Locations (1):
- Dept. of Oncology,The First Affiliated Hospital of Anhui Medical Univesrsity, Hefei, Anhui, China